CLINICAL TRIAL: NCT05469243
Title: A Retrospective Study Determine the Impact of Psychedelic Therapy for Dimensional Measures of Wellness
Brief Title: Psychedelic Therapy for Wellness Studies Retrospectively
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Canadian Forces Health Services Centre Ottawa (Other)
Responsible Party: Principal Investigator, Gaurav Gupta, Principal Investigator, Canadian Forces Health Services Centre Ottawa
Other Study IDs: 2022-013
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Well Aging
Keywords: wellness; psychedelics
MeSH Terms: interventions — Hallucinogens

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- psychedelics: 50 non active military participants not under the care of Dr. Gupta will be recruited through word of mouth and advertising to self-identify as having used psychedelic medicine for non recreational purposes (Appendix B recruitment letter). In addition to demographic information, they will be asked to complete the PGIC and anxiety, mood, pain and disability subscales, PEG, HADS and DI, provide information on their past medical history, nature/indications for use, and adverse events. This data will be collected once per participant and they will be able to speak with a research associate if further clarification if necessary at anytime.
  Interventions: Drug: Psychedelic

INTERVENTIONS:
Drug: Psychedelic — retrospective survey of previous use

SUMMARY:
The overall aim of this study is to assess the efficacy psychedelics for improving measures of wellness using a retrospective, single period, cohort study

DETAILED DESCRIPTION:
Previous research has largely focused on treating specific diagnostics groups such as depression, chronic pain, anxiety disorders with various approaches. With the significant overlap in symptomology with respect to diagnostic criteria and the presence of comorbidity, the results are challenging to extrapolate to real world applications. Therefore many authors have argued relying less on specific diagnoses, and instead focus on wellness, where symptom clusters or so called dimensions are explored independently.

The WHO constitution states: "Health is a state of complete physical, mental and social well-being and not merely the absence of disease or infirmity." An important implication of this definition is that health is more than just the absence of disorders or disabilities. Health is a state of well-being in which an individual realizes his or her own abilities, can cope with the normal stresses of life, can work productively and is able to contribute to his or her community.

Research Objective: In the current research investigators seek to measure the self-reported treatment effects of psychedelics (Psilocybin, 3,4-Methylenedioxymethamphetamine, N,N-Dimethyltryptamine, Lysergic Acid Diethylamide and Ketamine) for non recreational purposes (i.e., to self-medicate to ameliorate symptoms of suffering). Investigators will use a composite score of patient global perception, along with pain, function and mood scores as the measure of wellness, an approach to measurement which has not been done to date. Investigators follow previous work in this area, using a patient retrospective self-report study design, allowing for a safe way to develop further evidence in this area of care.

Participants and Procedure: 50 non active military participants not under the care of Dr. Gupta will be recruited through word of mouth and advertising to self-identify as having used psychedelic medicine for non recreational purposes (Appendix B recruitment letter). In addition to demographic information, they will be asked to complete the PGIC and anxiety, mood, pain and disability subscales, PEG, HADS and DI, provide information on their past medical history, nature/indications for use, and adverse events. This data will be collected once per participant and they will be able to speak with a research associate if further clarification if necessary at anytime.

Risks and Risk Mitigation: Participation in this study is voluntary and volunteers can withdraw consent at any time or skip any question they would prefer not to answer without having any effect on access to future medical care. Due to the nature of this study there are no additional associated risks. Patients can ask to be contacted by the research team should they wish to discuss any concerns, but will be apprised that this will breach their anonymity.

The PI agree to maintain accurate and secure records. The spreadsheet generated from this data will be password protected and anonymized. Only the research team will have access to this data and no patients will be identifiable unless they provide contact information requesting follow up.

Benefits and Military Significance: Outcomes of this project could potentially improve the quality of care for patients with various types of suffering by providing initial insights into these emerging treatments. The Canadian Forces specifically has considerably high rates of patients with comorbid pain and mental health issues. Therefore determining the impact on wellness could lead to further validation of treatments to improve quality of life, personal and occupational function.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 - 99
2. Self-report of past psychedelic medicine use for therapeutic purposes in the last 3 years
3. While a consent letter will be provided, patients will only be asked to agree to the terms without providing their names (i.e., unsigned consent procedures) given the potential legal ramifications of identification
4. Civilian or military veterans.

Exclusion Criteria:

1. Past psychedelic medicine use for non- therapeutic purposes
2. Only the most recent experience will be commented on
3. Active Military Members
4. Given the retrospective nature of the trial no other exclusion criteria outside not meeting the inclusion criteria are necessary.
5. In general patient participation will be anonymous given that access to medication may not have been considered legal. However in cases where there are concerns about a serious health issues and the patient can be identified, they will be to ensure appropriate follow up can be arranged.

Ages: 19 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — man, woman, other
Study Population: 50 non active military participants not under the care of Dr. Gaurav Gupta will be recruited. Colleagues will be informed that have may patients that could be candidates, in addition to advertising on a website and social media (eg facebook, instragram and/or twitter). The catchment will be set to Canada but will be expanded if the recruitment fails. Participants will therefore self-identify as having used psychedelic medicine for non recreational purposes (Appendix B recruitment letter).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2025-08-18 (Estimated); Study Completion 2025-08-27 (Estimated)

PRIMARY OUTCOMES:
patient's global impression of change | retrospective used in last 3 years
  patient's global impression of change (PGIC) has been used to estimate clinical change with a score of at least (moderate/much better), will be considered the minimally important clinically important difference. Scores 1-7 with higher scores associated with better outcome.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | baseline (current)
  The Hospital Anxiety and Depression Scale (HADS) is used to measure anxiety and depression in a general medical population of patients. The questionnaire comprises seven questions for anxiety and seven questions for depression interspersed within the questionnaire and scored separately. High scores note higher severity of illness.
Pain, Enjoyment and General Activity Scale (PEG) | baseline (current)
  Pain, Enjoyment and General Activity Scale (PEG) which is a 3-question scale with scores from 0-10 for each (total 30) looking to describe the change (if any) in activity limitations, symptoms, emotions and overall quality of life, related to the pain condition. Higher scores indicate poorer pain and function.
The Disability Index (DI) | baseline (current)
  7-item questionnaire adapted from the pain disability index to investigate the magnitude of self-reported related disability, independent of diagnosis. The items of the questionnaire are assessed on a 0-10 numeric rating scale in which 0 means no disability and 10 is maximum disability. (max score 70)

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Gupta, Principal Investigator — GG MPC
Locations (1):
- Gaurav Gupta MPC, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No